CLINICAL TRIAL: NCT04278547
Title: Phase IV Clinical Trial, Open, Randomized, Controlled and Multicentric, With Two Parallel Groups, to Assess the Efficacy of a Preventive Strategy Against Cytomegalovirus Infection in Heart Transplant Patients, Based on the Specific Basal T Cell Response Against Cytomegalovirus: ELISPOT-TC
Brief Title: Multicenter Clinical Trial to Evaluate the Efficacy of a Preventive Strategy Against CMV Infection in Heart Transplant Patients, Based on the Specific T Cells Response
Acronym: ELISPOT-TC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Elena García Romero, Elena García Romero, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI19/01610
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Heart Transplant Infection; CMV Infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Intervention Model Description: Phase IV clinical trial (with authorized treatment), randomized (2:1), controlled, open label and multicentric, with two parallel groups (Experimental group: preventive strategy based on the ELISPOT IFN-γ result: If patients are stratified as high risk they will receive prophylaxis with valgancyclovir for 3 months and if they are stratified as low risk they will be treated with preemptive therapy guided by CMV polymerase chain reaction analysis; Control group: Standard of care, universal prophylaxis with valgancyclovir for 3 months).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Preventive strategy based on the ELISPOT IFN-γ result: If patients are stratified as high risk they will receive prophylaxis with valgancyclovir for 3 months and if they are stratified as low risk they will be treated with preemptive therapy guided by CMV polymerase chain reaction analysis;
  Interventions: Diagnostic Test: ELISPOT IFN-γ assay
- Control group (No Intervention): Standard of care, universal prophylaxis with valgancyclovir for 3 months).

INTERVENTIONS:
Diagnostic Test: ELISPOT IFN-γ assay — ELISPOT IFN-γ diagnostic test: Evaluation of specific cellular immune response against the IE-1 antigen and the CMV pp65, using the technique ELISPOT IFN-γ and individualize the preventive strategy according to the result. In patients with a ELISPOT of "low risk" will be made advance therapy (preemptive therapy) guided by PCR of CMV In patients with a "high risk" ELISPOT, universal prophylaxis with valganciclovir will be performed oral (900 mg / 24h) or intravenous ganciclovir (5-10 mg / Kd / day) in case the oral route is not available.
  Other Names: Valganciclovir
  Arms: Experimental group

SUMMARY:
This study evaluates the efficacy and safety of an individualized preventive strategy against CMV infection in CMV seropositive heart transplant patients based on the specific basal response of the lymphocytes againts CMV (ELISPOT Interferon-γ assay).

In two thirds of the patients a preventive strategy will be carried out based on the result of the ELISPOT IFN-γ assay and in one third of the patients the standard of care strategy will be carried out (universal prophylaxis).

DETAILED DESCRIPTION:
Background: The prevention of Cytomegalovirus (CMV) infection in cardiac transplant patients is currently based exclusively on the performance of the serotypes of the receptor and the donor. Despite prophylactic treatment with valganciclovir or preemptive therapy through serial monitoring of blood viral copies, the rate of infection or CMV disease remains high and has a negative clinical impact. The evaluation of the specific T lymphocytes cellular immune response against 2 CMV antigens prior to kidney transplantaction, using the ELISPOT IFN-γ assay discriminates in a better way which patients will develop CMV infection.

Objetives: To compare the cumulative incidence of CMV infection during the first year post-heart transplant amongst CMV seropositive recipients in 12 national centers, where the prophylactic strategy regarding CMV infection will be guided by the ELISPOT IFN-γ assay or not (control). Main variable: number of patients who have CMV infection in the first year post-trasplant (HT).

Hyphotesis: A preventive strategy against CMV infection in CMV seropositive heart transplant patients, based on the specific basal response of the T lymphocytes against CMV, ELISPOT IFN-γ assay, is effective, safe and not inferior than the control group in terms of infection CMV rates. Design: The investigators propose a phase IV clinical trial (with authorized treatment), randomized (2:1), controlled, open label and multicentric, with two parallel groups (Experimental group: preventive strategy based on the ELISPOT IFN-γ result: If patients are stratified as high risk they will receive prophylaxis with valgancyclovir for 3 months and if they are stratified as low risk they will be treated with preemptive therapy guided by CMV polymerase chain reaction analysis; Control group: Standard of care, universal prophylaxis with valgancyclovir for 3 months).

Follow-up: 1 year. Duration of the trial: 3 years. Sample size: 188 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or more), both sexes, heart transplant patients.
* Patients with positive IgG against CMV (seropositive).
* Informed consent given by the subject or his legal representative.
* Availability of obtaining recipient and donor serologies.
* Availability of obtaining biological samples of peripheral blood post-transplant to be able to perform the ELISPOT IFN-γ assay.
* Women of childbearing age who use effective contraceptive measures during and until, so less, 30 days after treatment. Men who use contraceptive measures of barrier during and for at least 90 days after treatment, unless there is certainty that the female partner does not run the risk of becoming pregnant.

Exclusion Criteria:

* Pregnancy and / or breastfeeding period.
* Patients with contraindication for the use of valganciclovir or ganciclovir.
* Patients receiving thymoglobulin as induction therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-03-25 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have CMV infection in the first year post heart transplant. | One year
  Any viremia

SECONDARY OUTCOMES:
Number of patients with late CMV infection. | One year
  Number of patients with late CMV infection who have received prophylaxis with valganciclovir or ganciclovir (group 1 a and control group), once the treatment is finished.
Number of patients with acute rejection. | One year
Number of patients with vascular graft disease. | One year
Number of patients with other bacterial or viral opportunistic infections. | One year
Number of patients with leukopenia secondary to prophylaxis. | One year
Number of patients with neutropenia secondary to prophylaxis. | One year
Number of leukopenia patients presenting with other bacterial infections or viral. | One year
Number of deceased patients during hospital admission post-heart transplant. | One year
Number of deceased patients, related to CMV infection, in the first year post-transplant. | One year
Number of deceased patients, related to CMV disease, in the first post-transplant year. | One year
Number of patients who died from any cause in the first year post-heart transplant. | One year
Title of specific Inmunoglobulin G antibodies against serum CMV. | One year
Title of nonspecific serum gammaglobulins. | One year
CMV-specific memory response B (ELISPOT B). | One year
Number of patients whose ELISPOT varies from low to intermediate or high risk. | One year
Number of patients whose ELISPOT varies from intermediate or high risk to low risk. | One year
Number of spots against the IE-1 antigen. | One year
Number of spots against the pp65 antigen. | One year
Number of copies of CMV DNA measured by polymerase chain reaction (PCR). | One year
Estimate the economic cost of both strategies studied in this clinical trial | One year

CONTACTS AND LOCATIONS:
Overall Officials: José González Costello, Principal Investigator — Cardiologist
Locations (1):
- Hospital Universitari de Bellvitge, Barcelona, Spain